CLINICAL TRIAL: NCT01610193
Title: The Value of Pancreatic Stone Protein in Predicting Acute Appendicitis in Patients Presenting at the Emergency Department With Abdominal Pain
Brief Title: The Value of Pancreatic Stone Protein in Predicting Acute Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Laikο General Hospital, Athens (Other); University of Athens (Other); Kantonsspital Münsterlingen (Other)
Responsible Party: Sponsor
Other Study IDs: PSP_Appendix
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Appendicitis; Abdominal Pain; Abdominal Sepsis
Keywords: Pancreatic Stone Protein; Abdominal pain; Acute appendicitis; Alvarado score; Appendectomy; Sensitivity and specificity
MeSH Terms: conditions — Appendicitis; Abdominal Pain; Intraabdominal Infections; Hypersensitivity | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum or plasma of 245 patients.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Right sided abdominal pain: Patients that present at the Emergency Department with abdominal pain and a clinical suspicion of appendicitis.
  Interventions: Procedure: Appendicectomy

INTERVENTIONS:
Procedure: Appendicectomy — Also known as appendectomy, surgical removal of the appendix. Laparoscopic (single or 4 port), McBurney's incision, mid-line laparotomy, laparoscopic converted to open.
  Other Names: Appendectomy or appendisectomy

SUMMARY:
PSP (Pancreatic Stone Protein) is a compound naturally produced mainly in the pancreas and the gut. There is evidence from experimental and clinical trials that the levels of PSP in the blood rise in the presence of inflammation or infection. What is not yet well known about PSP is whether it is superior to other established blood tests (e.g. WBC or CRP) in predicting appendicitis in patients that present at the emergency room with abdominal pain and a clinical suspicion of appendicitis.

DETAILED DESCRIPTION:
Interim analysis will be performed once 123 patients are recruited. A power analysis will be performed and the sample size re-calculated based on the actual and precise data collected. At interim analysis, the external data monitoring committee will decide upon the continuation or discontinuation of the trial, as well the potential need to modify the sample size. If any changes are suggested by the external data monitoring committee, the principal investigators will decide on the feasibility of the potential changes and submit a formal addendum to the ethics committee. No changes will be made to the protocol or study design unless first approved by the ethics committee. Any changes to the protocol approved by the ethics committee will be updated at clinicaltrials.gov

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age (subject to the current ethics approval protocol, may change)
* Clinical suspicion of appendicitis as the primary or differential diagnoses
* Patients able to provide informed consent

Exclusion Criteria:

* Age <18 years of age (subject to the current ethics approval protocol, may change)
* Abdominal discomfort without tenderness or rebound or clinical suspicion of appendicitis
* Pregnancy
* Patients with impaired consciousness
* Patients not able to provide informed consent
* Patients that will receive an appendicectomy as part of another elective procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that will present at the emergency department with abdominal pain and a clinical suspicion of acute appendicitis.
Sampling Method: Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of PSP in diagnosing appendicitis | 1 day
  ROC Curve analysis and predictive value of PSP (Pancreatic Stone Protein) in diagnosing appendicitis

SECONDARY OUTCOMES:
Accuracy of CRP in diagnosing appendicitis | 1 day
  ROC Curve analysis and predictive value of CRP (C-Reactive Protein) in diagnosing appendicitis
Accuracy of WCC in diagnosing appendicitis | 1 day
  ROC Curve analysis and predictive value of WCC (White Cell Count) in diagnosing appendicitis
Accuracy of the "Alvarado Score" in diagnosis appendicitis | 1 day
  ROC Curve analysis and predictive value of Alvarado Score in diagnosing appendicitis
Accuracy of USS in diagnosing appendicitis | 1 day
  ROC Curve analysis and predictive value of Ultrasound Scanning (USS) in diagnosing appendicitis, most commonly performed in young females
Accuracy of CT in diagnosing appendicitis | 1 day
  ROC Curve analysis and predictive value of CT (Computer Tomography) in diagnosing appendicitis, most commonly performed in the elderly

OTHER OUTCOMES:
Independent predictors of appendicitis | 1 day
  Multivariate analysis of to identify independent clinical, laboratory and imaging predictors of appendicitis

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri A Raptis, MD, MSc, Principal Investigator — University Hospital Zurich, Department of Surgery; Rolf Graf, PhD, Study Chair — University Hospital Zurich, Department of Surgery
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Zurich, Canton of Zurich
  - University Hospital Zurich, Department of Surgery, Zurich

REFERENCES:
- [Background] Alvarado A. A practical score for the early diagnosis of acute appendicitis. Ann Emerg Med. 1986 May;15(5):557-64. doi: 10.1016/s0196-0644(86)80993-3. PMID 3963537
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Boeck L, Graf R, Eggimann P, Pargger H, Raptis DA, Smyrnios N, Thakkar N, Siegemund M, Rakic J, Tamm M, Stolz D. Pancreatic stone protein: a marker of organ failure and outcome in ventilator-associated pneumonia. Chest. 2011 Oct;140(4):925-932. doi: 10.1378/chest.11-0018. Epub 2011 Aug 11. PMID 21835904
- [Background] Keel M, Harter L, Reding T, Sun LK, Hersberger M, Seifert B, Bimmler D, Graf R. Pancreatic stone protein is highly increased during posttraumatic sepsis and activates neutrophil granulocytes. Crit Care Med. 2009 May;37(5):1642-8. doi: 10.1097/CCM.0b013e31819da7d6. PMID 19325491
- [Background] Graf R, Schiesser M, Reding T, Appenzeller P, Sun LK, Fortunato F, Perren A, Bimmler D. Exocrine meets endocrine: pancreatic stone protein and regenerating protein--two sides of the same coin. J Surg Res. 2006 Jun 15;133(2):113-20. doi: 10.1016/j.jss.2005.09.030. Epub 2005 Dec 19. PMID 16360171
- [Background] Bimmler D, Graf R, Scheele GA, Frick TW. Pancreatic stone protein (lithostathine), a physiologically relevant pancreatic calcium carbonate crystal inhibitor? J Biol Chem. 1997 Jan 31;272(5):3073-82. doi: 10.1074/jbc.272.5.3073. PMID 9006958
- [Background] Planas R, Pujol-Autonell I, Ruiz E, Montraveta M, Cabre E, Lucas-Martin A, Pujol-Borrell R, Martinez-Caceres E, Vives-Pi M. Regenerating gene Ialpha is a biomarker for diagnosis and monitoring of celiac disease: a preliminary study. Transl Res. 2011 Sep;158(3):140-5. doi: 10.1016/j.trsl.2011.04.004. Epub 2011 May 30. PMID 21867979
- [Background] Jin CX, Hayakawa T, Ko SB, Ishiguro H, Kitagawa M. Pancreatic stone protein/regenerating protein family in pancreatic and gastrointestinal diseases. Intern Med. 2011;50(15):1507-16. doi: 10.2169/internalmedicine.50.5362. Epub 2011 Aug 1. PMID 21804274
- [Derived] Tschuor C, Raptis DA, Limani P, Bachler T, Oberkofler CE, Breitenstein S, Graf R. The value of pancreatic stone protein in predicting acute appendicitis in patients presenting at the emergency department with abdominal pain. BMC Gastroenterol. 2012 Oct 25;12:154. doi: 10.1186/1471-230X-12-154. PMID 23098130